CLINICAL TRIAL: NCT03755700
Title: Antioxidants for Preventing Contrast-Induced Acute Kidney Injury After Coronary Artery Catheterization
Brief Title: Vitamin E and N-acetylcysteine for Preventing Contrast-Induced Acute Kidney Injury After Coronary Artery Catheterization
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rajaie Cardiovascular Medical and Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Intervention-01
Record Dates: First submitted 2018-11-25; First posted 2018-11-28 (Actual); Last update posted 2018-11-30 (Actual); Status verified 2018-11

CONDITIONS: Coronary Artery Disease; Coronary Artery Angiography; Coronary Catheterization; Contrast-induced Nephropathy; Stable Angina; Acute Coronary Syndrome
MeSH Terms: conditions — Coronary Artery Disease; Angina, Stable; Acute Coronary Syndrome | interventions — Vitamin E; Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Normal saline 0.9% infusions (1 mL/kg) for 12 hours prior to and after coronary catheterization combined with the placebos of both vitamin E and NAC (i.e. the placebo of vitamin E as a soft gel capsule and the placebo of NAC as an effervescent tablets along with a glass of water with the same consumption order used in the groups 2 and 3, respectively).
  Interventions: Drug: Placebo oral capsule; Drug: Placebos; Drug: Normal Saline Flush, 0.9% Injectable Solution
- Vitamin E (Active Comparator): Normal saline 0.9% infusions (1 mL/kg) for 12 hours prior to and after coronary catheterization combined with vitamin E 800 IU orally 2 hours before intervention and 400 IU orally 4 hours after intervention plus the placebo of NAC with a consumption order similar to group 3.
  Interventions: Drug: Vitamin E; Drug: Placebos; Drug: Normal Saline Flush, 0.9% Injectable Solution
- NAC (Active Comparator): Normal saline 0.9% infusions (1 mL/kg) for 12 hours prior to and after coronary catheterization combined with NAC 1200 mg orally 2 hours before intervention and 1200 mg orally 4 hours after intervention plus the placebo of vitamin E with the consumption order similar to group 2.
  Interventions: Drug: N-acetyl cysteine; Drug: Placebo oral capsule; Drug: Normal Saline Flush, 0.9% Injectable Solution

INTERVENTIONS:
Drug: Vitamin E — As a gel capsule of vitamin E 800 IU orally 2 hours before intervention and 400 IU orally 4 hours after intervention
  Arms: Vitamin E
Drug: N-acetyl cysteine — As an effervescent tablets of NAC 1200 mg orally 2 hours before intervention and 1200 mg orally 4 hours after intervention
  Arms: NAC
Drug: Placebo oral capsule — The placebo of vitamin E as a soft gel capsule with the consumption order similar to vitamin e group
  Arms: NAC; Placebo
Drug: Placebos — The placebo of n-acetylcysteine as a tablet with the consumption order similar to n-acetylcysteine group
  Arms: Placebo; Vitamin E
Drug: Normal Saline Flush, 0.9% Injectable Solution — Normal saline 0.9% infusions (1 mL/kg) for 12 hours prior to and after coronary catheterization

SUMMARY:
In a double-blinded randomized clinical trial, all patients undergoing coronary artery catheterization who will met our criteria, will be enrolled into three groups to receive either, vitamin e, n-acetylcysteine, or placebo. The aim of study will be to compare the superiority of vitamin e over n-acetylcysteine for the prevention of contrast-induced acute kidney injury (CIAKI).

DETAILED DESCRIPTION:
Patients aged ≥18 years with chronic kidney disease who undergo coronary catheterization will be enrolled into the study if they meet the inclusion criteria. Patients will be randomly assigned into three groups in a 1:1:1 ratio (Computer-generated random number will be used to assign a patient in either group): we will use simple randomization for assigning each patient in a group. The participants, physicians and outcome assessors will be blinded throughout the trial until the opening of the randomization cold.

All patients will be entered into three group and they will be given normal saline 0.9%, vitamin E, NAC, and the placebos of both regimens. The vitamin E will be given as a soft gel capsule and its placebo will have the same shape and taste. The NAC will be given as an effervescent tablet with a glass of water for consumption and its placebo will also have the same shape and taste. These drugs will be given in addition to the routine hydration therapy which will be given to all patients.

Primary outcome will be the development of CIAKI. Secondary outcomes will be the development of major adverse cardiovascular events and any events till evaluating the CIAKI within 48-72 hours after intervention.

ELIGIBILITY:
Inclusion Criteria:

Patients aged ≥18 years with baseline estimated glomerular filtration rate (eGFR) <60 mL/min per 1.73 m2 (based on the Modification of Diet in Renal Disease study group formula) who undergo coronary catheterization (i.e. coronary angiography and percutaneous coronary intervention [PCI]) will be invited to the study if they meet the inclusion criteria: stable angina with ischemia and indication for coronary angiography, non-ST-segment elevation (NSTE) acute coronary syndrome (ACS) requiring an early invasive strategy, and patients undergoing elective PCI .

Exclusion Criteria:

acute ST-segment elevation myocardial infarction, high-risk NSTE-ACS warranting emergency coronary angiography (<2 hours), cardiogenic shock, pulmonary edema, overt heart failure and/or ejection fraction <30%, ACS undergoing coronary angiography or angioplasty during the previous 5 days, sensitivity to contrast medium, recent administration of contrast medium for any reason, AKI, history of dialysis, pregnancy, newly prescribed angiotensin converting enzyme inhibitors or angiotensin receptor blockers, bleeding and/or coagulopathy diseases, and consumption of nephrotoxic drugs, vitamin E, vitamin C, or N-acetylcysteine (NAC) at least 48 hours before intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Contrast-induced acute kidney injury | 48 to 72 hours after coronary catheterization
  Contrast-induced acute kidney injury defined as an absolute increase ≥0.5 mg/dL or a relative increase ≥25% over baseline serum creatinine concentration within 48-72 hours after administration of contrast media.

SECONDARY OUTCOMES:
Changes in the levels of serum creatinine | 48-72 hours post-procedure
  Changes in serum creatinine after coronary artery catheterization
eGFR within 48-72 hours after coronary catheterization | 48-72 hours post-procedure
  Changes in eGFR after coronary artery catheterization
Changes in complete blood cell count components from baseline to follow-up | 48-72 hours post-procedure
  Changes in complete blood cell count components after coronary artery catheterization
Length of hospital stay | 48-72 hours post-procedure
  Length of hospital stay
Requirement for renal replacement therapies | 48-72 hours post-procedure
  Requirement for renal replacement therapies, ie, any kind of dialysis or renal transplantation
Post-procedure acute coronary syndrome (ACS) events | 48-72 hours post-procedure
  Recurrent acute coronary syndrome after coronary artery catheterization
Post-procedure cerebrovascular events | 48-72 hours post-procedure
  Cerebrovascular events after coronary artery catheterization
In-hospital mortality | 48-72 hours post-procedure
  In-hospital mortality after coronary artery catheterization
Post-procedure atrial fibrillation | 48-72 hours post-procedure
  Atrial fibrillation after coronary artery catheterization
Post-procedure bleeding | 48-72 hours post-procedure
  Bleeding events after coronary artery catheterization
Pulmonary embolism | 48-72 hours post-procedure
  Pulmonary embolism after coronary artery catheterization
Re-intervention | 48-72 hours post-procedure
  Repeated coronary artery catheterization

CONTACTS AND LOCATIONS:
Locations (1):
- Rajaie cardiovascular medical and research center, Tehran, Iran

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rezaei Y, Khademvatani K, Rahimi B, Khoshfetrat M, Arjmand N, Seyyed-Mohammadzad MH. Short-Term High-Dose Vitamin E to Prevent Contrast Medium-Induced Acute Kidney Injury in Patients With Chronic Kidney Disease Undergoing Elective Coronary Angiography: A Randomized Placebo-Controlled Trial. J Am Heart Assoc. 2016 Mar 15;5(3):e002919. doi: 10.1161/JAHA.115.002919. PMID 27068631
- [Background] Rezaei Y, Hemila H. Vitamins E and C May Differ in Their Effect on Contrast-Induced Acute Kidney Injury. Am J Kidney Dis. 2017 May;69(5):708-709. doi: 10.1053/j.ajkd.2016.12.022. Epub 2017 Mar 6. No abstract available. PMID 28279510